CLINICAL TRIAL: NCT07307365
Title: Evaluation of the Clinical Performance of the PremaSure Kit to Assess Premature Delivery Risk in Symptomatic Pregnant Patients
Status: Recruiting | Type: Observational
Sponsor: Rea Diagnostics SA (Industry)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Other Study IDs: REA-2024-02260
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Preterm Delivery
Keywords: Preterm Delivery; Self-test
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to determine the clinical performance of the PremaSure kit, more precisely to assess whether the PremaSure kit can be used as a self-test to assess the risk of premature delivery in patients showing symptoms of premature delivery. The sensitivity and specificity of the test will be determined using as an outcome the delivery of the patient in the 7/14 days following the test.

The simplified procedure is the following:

1. Patients are recruited and screened for eligibility criteria
2. A healthcare professional collects a vaginal swab from the patient
3. The collected sample is tested on the PremaSure kit
4. Pregnancy outcome is compared to the PremaSure kit's result

DETAILED DESCRIPTION:
Introduction:

Preterm birth is the first cause of death of infants below five years old. One of the key strategies to save preterm babies is to effectively identify women at risk of preterm birth. While current solutions for the assessment of prematurity risk rely on invasive examination performed by medical professional, the PremaSure is intended to be used by lay user, empowering them with a tool to monitor their pregnancy.

Measurement and procedures:

Consenting patient meeting all the inclusion and none of the exclusion critera will be swabbed by a healthcare professional to collect vaginal secretions. A study nurse will perform the test per the test's IFU. Information related to the patient's delivery will be collected after term to evaluate the predictive performance of the PremaSure kit.

Withdrawal and discontinuation:

Participants can withdraw their consent from the study at any time with no consequence for their clinical management. Patients do not have to provide any reason for withdrawing their consent. Patients who wish to withdraw consent for participation in the study, must notify the Principal Investigator by sending an email to or calling the Principal Investigator using the email address/ phone number mentioned in the ICF. Upon receipt of a notification that a patient wishes to withdraw from the study, the Principal Investigator will document the withdrawal in the eCRF and inquire whether the patient consents that already collected data can be kept on record.

Labelling of the device under investigation:

As the IVD device is not commercially available, the labelling shall indicate that the IVD device under investigation is exclusively for use in a performance study. Each device will have a unique identifying number to trace its origin and manufacturing lot.

Accountability of the IVD device:

Upon receipt at the study sites, the kits shall be stored in a secured location and only accessible for team members involved in the study.

Unused, expired or malfunctioning IVD devices shall be returned to the sponsor.

Monitoring plan:

For each of the sub-studies, a separate site initiation visit will be performed after all required approvals are obtained. As part of this visit the staff involved in the study at the study site will be trained on the procedures presented in this protocol. The devices/kits will be shipped to the site after authorization of the study by the Ethics Committee and approval of the required essential documents.

During the study, the monitor will contact and visit the site regularly. The monitor must have access, with reasonable prior notice, to the facilities of the study site and all source documents needed to verify adherence to the protocol as well as the completeness, consistency and accuracy of the data being entered on the eCRFs and other protocol-related documents. Additional checks of the consistency of the source data with the eCRFs will be performed according to the study-specific monitoring plan. The frequency of the monitoring visits will be mainly based on subject recruitment.

The investigator/delegate must ensure that the eCRFs are completed per the eCRF completion guidelines and that all requested subject files (e.g., ICF, medical notes/charts, other documentation verifying the activities conducted at the study) are available for review by the monitor. The required site staff must be available during the monitoring visits and allow necessary time to meet with the monitor to discuss study-related topics and issues.

A close-out visit will be performed for any initiated site.

Data recording:

Electronic Data Capture (EDC) will be used to collect eCRF data. The eCRF, based on RedCap solution, must be completed in a timely manner as per the eCRF completion guidelines.

The principal investigator and delegate site staff member(s) will be trained to enter and edit the data via a secure network, with secure access features (username, password and identification). While entering the data, the principal investigator/delegate will be instantly alerted to data queries by validated programmed checks. Additional review will be performed by the sponsor/monitor on an ongoing basis to check for unexpected patterns in data and for study monitoring. Should discrepant data be detected, a manual query will be issued for clarification of the data. The query will be visible to the principal investigator/delegate via the eCRF. Response/correction by the principal investigator/delegate will be performed directly in the eCRF. All eCRF entered data require must have documented background data which will remain available for the monitor and to health authorities queries and inspections. A complete electronic audit trail will be maintained in the EDC system. The investigator/delegate will approve the data, confirming its accuracy and completion by signing the eCRF electronically (as per US 21 CFR part 11). Data will be stored on secured servers in Switzerland.

Source data verification will be performed by the monitor. In the electronic database the sponsor shall have access to coded data that can be used to monitor patient recruitment and endpoint assessment.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Female patients above 18 years
* Gestational week from 22w+0 days to 35w+6 days
* Symptoms of prematurity.

Exclusion Criteria:

* Subject lacking capacity to provide informed consent
* Enrolment of the project leader, their family members, employees and other dependent persons
* Patients with ruptured amniotic membranes or blood in their vaginal discharge
* Patients with vaginal examination in the last 24 hours
* Previous enrolment in the current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological female can be included in the study.
Study Population: Pregnant patients with symptoms of premature delivery.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the clinical performance of the PremaSure kit | From enrollment to the delivery of the patient
  On the population of patients who have fully completed the study without experiencing a non-spontaneous delivery up to 14 days after the sample collection, we will determine the sensitivity, specificity, accuracy, positive and negative predictive values (PPV and NPV respectively) of the PremaSure test for the identification of pregnant women at risk of pre-term delivery at 7 and 14 days, respectively

SECONDARY OUTCOMES:
Estimation of the clinical performance of the PremaSure kit on sub-group population | From enrollment until the delivery of the patient
  Estimation of sensitivity and specificity, PPV, NPV and prevalence for the risk of pre-term delivery of sub-groups, defined as any combination of the categories derived from the pregnancy information collected in the context of the present study. The statistical study power may not be attained for each subgroup. The aforementioned values will be determined considering as an outcome a delivery at 7 days, 14 days, or at any duration following the test.
Estimation of correlation coefficients between the participant pregnancy information and the outcome of the pregnancy | From enrollment until delivery of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universtaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland